CLINICAL TRIAL: NCT03389841
Title: Home Care for the Patient With Heart Failure: Can Caregiver Education Prevent Hospital Admissions? A Clinical Randomized Trial.
Brief Title: Home Care for the Patient With Heart Failure: Can Caregiver Education Prevent Hospital Admissions?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Stella Padula (Other)
Collaborators: University of Modena and Reggio Emilia (Other); Local Health Authority of Modena (Unknown)
Responsible Party: Sponsor-Investigator, Maria Stella Padula, local manager of the province of Modena, Italian College of General Practitioners
Organization: Italian College of General Practitioners (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MSP_01
Record Dates: First submitted 2017-12-27; First posted 2018-01-04 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure
Keywords: home care services; comorbidity; heart failure; caregivers; health education; patient admission
MeSH Terms: conditions — Heart Failure; Health Education | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Education of the caregiver
  Interventions: Other: Education
- No intervention (No Intervention): Usual care

INTERVENTIONS:
Other: Education — Education of the caregiver about early symptoms and signs of heart failure
  Arms: Intervention

SUMMARY:
The study is aimed to evaluate if the education of the caregiver is able to reduce hospital admissions of patients with heart failure assisted at home.

DETAILED DESCRIPTION:
The primary objective of the study is to assess whether an educational intervention aimed at increasing the caregiver's skills is able to reduce hospital admissions for any cause in patients with heart failure assisted at home.

The General Practitioners who agree to participate are randomized in two groups: a) intervention group, whose patients are assisted in accordance with the procedures established by the project; b) control group, whose patients continue to be assisted in the usual modality.

The intervention consists of an educational session for each caregiver aimed at improving his ability to recognize early symptoms and signs of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* adults of any age and gender in NYHA (New York Heart Association) classes II, III, IV, assisted exclusively at home;
* willingness and ability to sign a written informed consent;
* presence of a person who cared for the patient in a prevalent and regular way;
* willingness of the caregiver to attend a training meeting.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-04-10 (Actual); Study Completion 2016-04-10 (Actual)

PRIMARY OUTCOMES:
Hospital admissions for any cause | Twelve months
  Hospital admissions for any cause

SECONDARY OUTCOMES:
Hospital admissions for cardiovascular causes | Twelve months
  Hospital admissions for cardiovascular causes
Mortality for general or cardiovascular causes | Twelve months
  Mortality for general or cardiovascular causes

IPD SHARING:
Plan to Share IPD: Yes
all Individual Participant Data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Padula MS, D'Ambrosio GG, Tocci M, D'Amico R, Banchelli F, Angeli L, Scarpa M, Capelli O, Cricelli C, Boriani G. Home care for heart failure: can caregiver education prevent hospital admissions? A randomized trial in primary care. J Cardiovasc Med (Hagerstown). 2019 Jan;20(1):30-38. doi: 10.2459/JCM.0000000000000722. PMID 30394960